CLINICAL TRIAL: NCT00367835
Title: A Double-Blind, Randomized, Multi-Center, Flexible Dose Study Evaluating the Efficacy and Safety of SPD503 (Guanfacine Hydrochloride) in Children Aged 6-12 With Symptoms of Oppositionality and a Diagnosis of Attention Deficit/Hyperactivity Disorder
Brief Title: SPD503 (Guanfacine Hydrochloride) in ADHD Plus Oppositional Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD503-307
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SPD503 (Guanfacine hydrochloride) (Experimental)
  Interventions: Drug: SPD503 (Guanfacine hydrochloride)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD503 (Guanfacine hydrochloride) — Subjects will start at 1mg tablet each morning and will subsequently be titrated (in 1 mg weekly increments) to optimal dose based upon tolerance and response to investigational product (not to exceed 4 mg/day).
  Arms: SPD503 (Guanfacine hydrochloride)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To assess efficacy and safety of SPD503(guanfacine hydrochloride) in subjects with ADHD and oppositional symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with ADHD and oppositional symptoms
* ADHD-RS>=24
* CGI >=4
* T-score of Opp subscale CPRS-R:L >=65
* Normal ECG and BP
* >= 55 lbs

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2006-12-04 (Actual); Primary Completion 2008-01-04 (Actual); Study Completion 2008-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (34):
- United States (34):
  - HOPE Research Institute, Phoenix, Arizona
  - Valley Clinical Research, El Centro, California
  - Peninsula Research Associates Inc, Rolling Hills Estates, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Amedica Research Institute, Inc, Hialeah, Florida
  - CORE Research, Inc, Maitland, Florida
  - Miami Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Childrens Developmental Center, Winter Park, Florida
  - Capstone Clinical Research, Libertyville, Illinois
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Pedia Research, Owensboro, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CRI Worldwide, LLC, Clementon, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester, School of Medicine and Dentistry, Rochester, New York
  - SUNY Upsate Medical University, Syracuse, New York
  - Piedmont Neuropsychiatry, Charlotte, North Carolina
  - Duke Child & Family Study Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Discovery and Wellness Center for Children, Cleveland, Ohio
  - BHI Inc, Moore, Oklahoma
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc, Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc, Salem, Oregon
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Claghorn-Lesem Research Clinic Inc, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - NeuroScience, Inc, Herndon, Virginia
  - Dominion Clinical Research, Midlothian, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington

REFERENCES:
- [Result] Connor DF, Findling RL, Kollins SH, Sallee F, Lopez FA, Lyne A, Tremblay G. Effects of guanfacine extended release on oppositional symptoms in children aged 6-12 years with attention-deficit hyperactivity disorder and oppositional symptoms: a randomized, double-blind, placebo-controlled trial. CNS Drugs. 2010 Sep;24(9):755-68. doi: 10.2165/11537790-000000000-00000. PMID 20806988
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html
- See also: FDA-approved label — http://www.intuniv.com/documents/INTUNIV_Full_Prescribing_Information.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 217 subjects were randomized (138 to SPD503 and 79 to placebo). However, only 214 subjects received at least one dose of study medication (136 for SPD503 and 78 for placebo). Therefore, 214 subjects constitute the safety population.
Groups:
- SPD503: Subjects will receive either 1, 2, 3, or 4 mg/day oral doses of SPD503 (Guanfacine hydrochloride)
Period: Overall Study
Arm/Group | SPD503 | Placebo
Started | 138 | 79
Completed | 109 | 48
Not Completed | 29 | 31
Not completed — Adverse Event | 14 | 1
Not completed — Protocol Violation | 1 | 7
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Lost to Follow-up | 1 | 4
Not completed — Lack of Efficacy | 3 | 12
Not completed — Subject in juvenile detention center | 1 | 0
Not completed — refused blood collection | 1 | 0
Not completed — Did not respond to calls | 1 | 0
Not completed — History of lead poisoning | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD503 | Placebo | Total
Number analyzed (Participants) | 138 | 79 | 217
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 138 | 79 | 217
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (1.73) | 9.3 (2.04) | 9.4 (1.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 19 | 69
  Male | 88 | 60 | 148
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 138 | 79 | 217

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Oppositional Subscale of the Conners' Parent Rating Scale-Revised Long Form (CPRS-R:L) Score at Up to 8 Weeks
Description: The oppositional subscale of the CPRS-R:L contains 10 items designed to reflect criteria for oppositional defiance disorder (ODD). Each item is scored on a range from 0 (not true at all) to 3 (very much true) with total scores ranging from 0 to 30. Higher scores are reflective of more severe symptoms.
Time Frame: Baseline and up to 8 weeks
Population: Full Analysis Set (FAS) defined as all randomized subjects who received at least one dose of any investigational product during this study and with a baseline and at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 130 | 75
Units on a scale | -10.8 (7.23) | -7.0 (7.63)
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS-IV) Total Score at Up to 8 Weeks
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and up to 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 130 | 75
Units on a scale | -23.8 (14.43) | -11.4 (12.65)
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

3. Secondary Outcome: Assessment of Clinical Global Impression-Severity of Illness (CGI-S)
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: up to 8 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 130 | 75
Participants
  1 (Normal, not at all ill) | 25 | 3
  2 (Borderline mentally ill) | 33 | 6
  3 (Mildly ill) | 29 | 15
  4 (Moderately ill) | 26 | 24
  5 (Markedly ill) | 13 | 22
  6 (Severely ill) | 4 | 5
  7 (Among the most extremely ill) | 0 | 0
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I)
Description: CGI-I consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: up to 8 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 130 | 75
Participants | 93 | 24
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Change From Baseline in the 40-Item Conduct Problem Scale of the New York Parent's Rating Scale-School-aged (NYPRS-S) Score at Up to 8 Weeks
Description: Each item on the NYPRS-S is scored from a range of 0 (not at all) to 3 (very much) with total scores ranging from 0 to 120. Higher scores are reflective of increased disease severity.
Time Frame: Baseline and up to 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 130 | 75
units on a scale | -15.6 (12.86) | -10.3 (13.25)
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Secondary Outcome: Change From Baseline in the Parent Stress Index-Short Form (PSI/SF) Score at Up to 8 Weeks
Description: The response to each of the 36 items on the PSI/SF is converted to a five-point scale from 1 (strongly agree) to 5 (strongly disagree) with total scores ranging from 36 to 180. A higher score is reflective of less stress for the parents.
Time Frame: Baseline and up to 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 109 | 57
Units on a scale | 17.3 (19.76) | 7.2 (18.29)
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA

7. Secondary Outcome: Number of Participants With Overall Satisfaction on the Medication Satisfaction Survey (MSS)
Description: The Medication Satisfaction Survey (MSS) consists of 11 questions each being answered with one of six responses (strongly agree, agree, somewhat agree, somewhat disagree, disagree, strongly disagree). Overall satisfaction with their child taking the study medication, Question #11, with a response of "strongly agree" or "agree".
Time Frame: up to 8 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 129 | 69
Participants | 84 | 21
Statistical Analysis 1: Comparison: SPD503 vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

8. Secondary Outcome: Change From Baseline in Electrocardiogram Results (QTcF Interval) at Up to 8 Weeks
Description: QTcF is the QT interval using Fridericia's correction formula. QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate (e.g., the faster the heart rate, the shorter the QT interval). The QT interval has to be corrected in order to aid interpretation.
Time Frame: Baseline and up to 8 weeks
Population: Safety population defined as all randomized subjects who received at least one dose of any investigational product during this study.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 107 | 58
msec | 5.2 (15.74) | 2.1 (17.41)

9. Secondary Outcome: Change From Baseline in Pulse Rate at Up to 8 Weeks
Time Frame: Baseline and up to 8 weeks
Population: Safety population
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 130 | 75
beats/min | -4.3 (11.89) | 0.7 (11.44)

10. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Up to 8 Weeks
Time Frame: Baseline and up to 8 weeks
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 130 | 75
mmHg | -2.6 (10.27) | 0.7 (8.18)

11. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Up to 8 Weeks
Time Frame: Baseline and up to 8 weeks
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SPD503 | Placebo
Number analyzed (Participants) | 130 | 75
mmHg | -1.3 (8.48) | 0.9 (7.38)

ADVERSE EVENTS:
Arm/Group | SPD503 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/78
Other Adverse Events (participants affected / at risk) | 115/136 | 47/78
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503 (N=136) | Placebo (N=78)
Somnolence (Nervous system disorders) | 69 | 5
Headache (Nervous system disorders) | 30 | 14
Sedation (Nervous system disorders) | 18 | 1
Dizziness (Nervous system disorders) | 7 | 3
Abdominal pain upper (Gastrointestinal disorders) | 16 | 2
Vomiting (Gastrointestinal disorders) | 10 | 5
Nausea (Gastrointestinal disorders) | 4 | 5
Fatigue (General disorders) | 15 | 4
Irritability (Psychiatric disorders) | 11 | 2
Affect lability (Psychiatric disorders) | 2 | 4
Blood pressure diastolic decreased (Investigations) | 8 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually